CLINICAL TRIAL: NCT05657483
Title: Inflammatory Index as a Predictor for Endometrial Cancer: an Observational Study
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Carlo Ronsini, Medical Doctor, University of Campania Luigi Vanvitelli
Other Study IDs: 0035563/i
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Neoplasms; Inflammatory Response
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial cancer patients: At least 18-year-old patients histologically diagnosed with endometrial cancer who will undergo surgical staging of disease after performing full-body CT-scan 30 days before the enrollment.
  Interventions: Diagnostic Test: Venous blood sample; Other: Surgical staging of endometrial cancer

INTERVENTIONS:
Diagnostic Test: Venous blood sample — Blood chemistry tests: neutrophil; lymphocyte; monocyte; platelet counts.
  Other Names: Blood chemistry test
Other: Surgical staging of endometrial cancer — Endometrial, adnexal, and lymphoid tissue samples.
  Other Names: Biopsy

SUMMARY:
It is a prospective observational trial. Primary goal is identification of an association between alteration of systemic inflammation indices, such as neutrophil-to-lymphocyte ratio (NLR), platelet-t- lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (MRL) and patients risk classification according to European Guidelines.

The population is represented by all women being admitted to the Gynecology Ward, through Emergency, who are affected by endometrial cancer. Participants will undergo surgery, and freely express their consent to participate in the study.

DETAILED DESCRIPTION:
Surgical treatment for endometrial cancer is class A radical hysterectomy according to Querleu-Morrow and bilateral adnexectomy with systematic pelvic lymphadenectomy. That allows the choice of adjuvant treatment, basing on anatomopathological risk information. Despite the standardization of adjuvant treatments, survival curves are heterogeneous in patients' responses. That is why European guide-lines have proposed a stratification of patients basing on oncological risk and molecular data (Microsatellite instability, aberrant P53, POLE gene mutation). The Investigators want to identify additional parameters to better define risk profiles. Systemic inflammation indices such as neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR) and lymphocyte-to-monocyte ratio (LMR) have shown prognostic value in several inflammatory conditions and solid tumors. Therefore, the Investigators have decided to explore their role also in recently diagnosed endometrial cancers, to find correlations with lymphovascular space invasion (LVSI), myometrial infiltration, histotype, and therefore with oncological risk classification. It is a prospective observational trial. Primary goal is identification of an association between alteration of systemic inflammation indices, such as neutrophil-to-lymphocyte ratio (NLR), platelet-t- lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (MRL) and patients risk classification according to European Guidelines.

The population is represented by all women being admitted to the Gynecology Ward, through Emergency, who are affected by endometrial cancer. Participants will undergo surgery, and freely express their consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically diagnosed with endometrial cancer.
* Patients undergoing surgical staging of the disease.
* Patients undergoing full-body CT-scan 30 days before enrollment.
* At least 18-year-old patients.

Exclusion Criteria:

* Unfit to plead.
* Patients with chronic inflammatory diseases (IBDs; rheumatic conditions).
* Synchronous tumors or cancer diagnosis in the previous 3 years.
* Patients undergoing steroid therapy in the last 30 days prior to recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with histological diagnosis of endometrial cancer undergoing surgical intervention who performed full-body CT-scan 30 days before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Grading | 30 days after surgery
  Anatomic pathology report of cell anaplasia in the sampled tumor
Staging | 30 days after surgery
  Anatomic pathology report of extent to which the cancer has spread
Histotype | 30 days after surgery
  Anatomic pathology report of tissue types that arise during the growth of cancer
Lymphovascular space invasion | 30 days after surgery
  Prognostic factor for recurrence and survival in endometrial cancer
Molecular profile | 30 days after surgery
  Biomarker testing of genes and/or proteins

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ronsini, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Università degli Studi della Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ronsini C, Iavarone I, Vastarella MG, Corte LD, Andreoli G, Bifulco G, Cobellis L, de Franciscis P. Additional Risk Factors Lead to a Measurable Inflammatory Response in Stage I Endometrial Cancer-A Prospective Multicentric Observational Study. Indian J Surg Oncol. 2025 Dec;16(6):1474-1481. doi: 10.1007/s13193-025-02228-5. Epub 2025 Feb 24. PMID 41415794